CLINICAL TRIAL: NCT03584503
Title: Effect of the Use of Endotracheal Tube With Subglottic Suction on Laryngospasm and Postoperative Complications in Rhinoplasty Operations
Brief Title: Effect of Use of Endotracheal Tube With Subglottic Suction in Rhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SACETT
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Rhinoplasty
Keywords: general anesthesia; laryngospasm; postoperative complications; rhinoplasty; Suction Above Cuff Endotracheal Tube
MeSH Terms: conditions — Laryngismus; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: A randomized prospective controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SA (Active Comparator): Group SA intubated with Suction Above Cuff Endotracheal Tube
  Interventions: Other: Suction Above Cuff Endotracheal Tube
- Group C (No Intervention): Group C intubated with classic endotracheal tube

INTERVENTIONS:
Other: Suction Above Cuff Endotracheal Tube — Suction Above Cuff Endotracheal Tube (SACETT) has a dorsal port above the cuff designed to allow continuous or intermittent suctioning of secretions from the subglottic space
  Arms: Group SA

SUMMARY:
Suction Above Cuff Endotracheal Tube (SACETT) has a dorsal port above the cuff designed to allow continuous or intermittent suctioning of secretions from the subglottic space. Thus, it facilitates suctioning of excessive secretions around the mouth and the cuff. In this study, we aimed to investigate the effect of the use of SACETT on laryngospasm and postoperative complications in rhinoplasty operations. This randomized controlled clinical trial was conducted in 132 patients undergoing rhinoplasty.

The investigators believe that the use of SACETT in rhinoplasty operations reduces the incidences of laryngospasm, emergence agitation, sore throat, swallowing difficulty, and PONV when compared with classic endotracheal tube.

DETAILED DESCRIPTION:
Suction Above Cuff Endotracheal Tube (SACETT) has a dorsal port above the cuff designed to allow continuous or intermittent suctioning of secretions from the subglottic space. Thus, it facilitates suctioning of excessive secretions around the mouth and the cuff. In this study, the investigators aimed to investigate the effect of the use of SACETT on laryngospasm and postoperative complications in rhinoplasty operations.

This randomized controlled clinical trial was conducted in 132 patients undergoing rhinoplasty. The patients were randomly divided into 2 groups: Suction Above Cuff Endotracheal Tube (n:66) (Group SA) and classic endotracheal tube (n:66) (Group C). Complications following general anesthesia were statistically analyzed among the two groups.

55 male patients and 77 female patients were included in the study. The incidences of postoperative laryngospasm and respiratory complications were found to be lower in Group SA compared to Group C. In addition, the incidences of agitation, postoperative nausea and vomiting (PONV), swallowing difficulty, and sore throat were found to be lower in Group SA compared to Group C. However, the incidences of cough, hypotension, and tachycardia were similar in both groups. No PONV, swallowing difficulty, and hypotension were observed in Group SA. The blood volume accumulated in the suction chamber was found to be greater in Group SA compared to Group C.

The investigators believe that the use of SACETT in rhinoplasty operations reduces the incidences of laryngospasm, emergence agitation, sore throat, swallowing difficulty, and PONV when compared with classic endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo rhinoplasty surgery,
* American Society of Anesthesiologists (ASA) I-II patients,
* Aged 18-65 years

Exclusion Criteria:

* Patients who had upper or lower respiratory tract infections,
* asthma,
* a history of allergy,
* who received isoflurane and desflurane for maintenance of anesthesia,
* who were the ASA class III-IV,
* and who had a long uvula,
* gastroesophageal reflux or sleep apnea,
* electrolyte disturbances such as hypomagnesemia and hypocalcemia,
* a BMI (body mass index) over 30 were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of laryngospasm | 1 mounth
  While the presence of findings such as apnea (an apneic event was counted by either documentation of apnea by nursing notes through visual observation or documented pauses ≥15 s), desaturation (peripheral oxygen saturation <85%) and inspiratory stridor (Stridor is a harsh, vibratory sound of variable pitch caused by partial obstruction of the respiratory passages that results in turbulent airflow through the airway) after extubation was considered as laryngospasm.

SECONDARY OUTCOMES:
emergence agitation | 1 mounth
  Riker Sedation-Agitation Scale Score ≥5 (7-Dangerous agitation: Pulling at endotracheal tube, trying to remove catheters, climbing over bedrail, striking at staff, thrashing side-to-side 6- Very agitated: Does not calm despite frequent verbal reminding of limits, requires physical restraints, biting endotracheal tube 5- Agitated: Anxious or mildly agitated, attempting to sit up, calms down on verbal instructions 4- Calm cooperative: Calm, easily arousable, follows commands 3- Sedated: Difficult to arouse, awakens to verbal stimuli or gentle shaking but drifts off again, follows simple commands 2- Very sedated: Arouses to physical stimuli but does not communicate or follow commands, may move spontaneously
  1- Unarousable: Minimal or no response to noxious stimuli, does not communicate or follow command)

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yüzkat, Assis prof, Study Chair — Yuzuncu Yil University
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mao Z, Gao L, Wang G, Liu C, Zhao Y, Gu W, Kang H, Zhou F. Subglottic secretion suction for preventing ventilator-associated pneumonia: an updated meta-analysis and trial sequential analysis. Crit Care. 2016 Oct 28;20(1):353. doi: 10.1186/s13054-016-1527-7. PMID 27788682
- [Result] Carter EL, Duguid A, Ercole A, Matta B, Burnstein RM, Veenith T. Strategies to prevent ventilation-associated pneumonia: the effect of cuff pressure monitoring techniques and tracheal tube type on aspiration of subglottic secretions: an in-vitro study. Eur J Anaesthesiol. 2014 Mar;31(3):166-71. doi: 10.1097/EJA.0000000000000009. PMID 24270899
- [Result] Alalami AA, Ayoub CM, Baraka AS. Laryngospasm: review of different prevention and treatment modalities. Paediatr Anaesth. 2008 Apr;18(4):281-8. doi: 10.1111/j.1460-9592.2008.02448.x. PMID 18315632
- [Derived] Yuzkat N, Demir CY. Effect of using the Suction Above Cuff Endotracheal Tube (SACETT) on postoperative respiratory complications in rhinoplasty: a randomized prospective controlled trial. Ther Clin Risk Manag. 2019 Apr 17;15:571-577. doi: 10.2147/TCRM.S200662. eCollection 2019. PMID 31114211